CLINICAL TRIAL: NCT05319587
Title: Phase 1/2 Study of Liposomal Annamycin in Combination With Cytarabine for the Treatment of Subjects With Acute Myeloid Leukemia (AML)
Brief Title: Study of Liposomal Annamycin in Combination With Cytarabine for the Treatment of Subjects With Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Moleculin Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MB-106; 2020-005493-10 (EudraCT Number)
Record Dates: First submitted 2022-02-22; First posted 2022-04-08 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Liposomal annamycin (Experimental)
  Interventions: Drug: Liposomal Annamycin; Drug: Cytarabine

INTERVENTIONS:
Drug: Liposomal Annamycin — 2-hour intravenous infusion liposomal annamycin daily for 3 consecutive days followed by 18 days off study drug (i.e., one treatment cycle = 21 days).
Drug: Cytarabine — Administered during cycle 1 at a dose of 2.0 g/m2/day by 4 hours IV infusion for 5 consecutive days and this dose will remain constant for all cohorts, including the expansion phase.

SUMMARY:
This is a Phase 1/2, multicenter, open-label, dose-escalation study that will determine the MTD and RP2D of L-Annamycin in combination with cytarabine for the treatment of subjects with AML.

DETAILED DESCRIPTION:
During Phase 1b, dose escalation will proceed according to a standard 3+3 design. An initial group of 3 subjects will be treated with an intravenous infusion of 190-mg/m2 L-Annamycin (Dose Level 1) for 3 consecutive days. Dose escalation will take place on the basis of safety assessments in sequential cohorts of 3 subjects each. Provided that there are no DLT's in the initial cohort of subjects treated at the 190 mg/m2/day dose level, the next cohort of subjects will receive the next highest L-Annamycin dose incremented by 40 mg/m2. In the absence of DLTs, dose escalation by 40 mg/m2 will continue in subsequent cohorts until an MTD is reached.

The dose and schedule of cytarabine during Cycle 1 (2.0 g/m2/day for 5 consecutive days) will remain constant for all cohorts. Enrolled subjects will receive cytarabine at a dose of 2.0 g/m2/day via intravenous infusion over 4 hours for 5 consecutive days (total dose cytarabine = 10.0 g/m2; starting on the first day of L-Annamycin treatment).

If no subject experiences a dose-limiting toxicity (DLT), based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5, which constitutes a study drug-related irreversible or not medically manageable Grade 3 or higher toxicity during the initial treatment through Day 28, the subsequent group of 3 subjects will receive the next higher L-Annamycin dose. However, if 1 of the 3 initial subjects experiences a DLT, the cohort of subjects at that dose level will be expanded to 6. If at least 2 of the 6 subjects experience a DLT, this will be considered a non-tolerated dose and the next 3 subjects will be treated at a lower dose. The dose of L-Annamycin will be de-escalated by 20- mg/m2/day. As such, if at least 2 out of 6 subjects receiving 230 mg/m2/day experience a DLT, the next 3 subjects will receive L-Annamycin at a dose of 210 mg/m2/day. If 1 of the 3 initial subjects experiences a DLT, the cohort of subjects will be expanded to 6 subjects. If at least 2 of the 6 subjects experience a DLT, this will be considered a toxic dose and the MTD will be the previously proven safe dose level (i.e., the next lowest dose level at which no DLTs occurred in a cohort of 3 subjects or at which fewer than 2 subjects in a cohort of 6 experienced a DLT).

In the expansion phase, up to 21 subjects will be enrolled at the MTD/RP2D to better define toxicity and evaluate efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has a pathologically confirmed diagnosis of AML by World Health Organization classification. This must be in the form of either a bone marrow aspirate or biopsy or a CBC that demonstrates >5% myeloblasts.
2. The subject has AML and has not received prior therapy or is refractory to or relapsed after induction therapy. To be defined as relapse, there must be >5% blasts in the bone marrow.
3. For the expansion phase only (i.e., after the MTD/RP2D is established), subjects must be treated with L-Annamycin as first- second- or third-line therapy (i.e., subjects will not have received more than two prior therapies).
4. The subject is age ≥18 years at the time of signing informed consent.
5. The subject has received no chemotherapy, radiation, or major surgery within 2 weeks prior to first dose of study drug and/or has recovered from the toxic side effects of that therapy unless treatment is indicated as a result of progressive disease, such as hydroxyurea.
6. The subject has received no investigational therapy within 4 weeks of the first dose of study drug.
7. The subject has an Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
8. The subject has adequate laboratory results including the following:

   1. Bilirubin ≤2 times the upper limit of normal unless due to Gilbert Syndrome or leukemic infiltration of the liver.
   2. Serum glutamic-oxaloacetic transaminase (SGOT), serum glutamic-pyruvic transaminase (SGPT), and alkaline phosphatase <2.5 times the upper limit of normal unless due to organ involvement.
   3. Adequate renal function with creatinine levels ≤2 times the upper limit of normal.
9. The subject can understand and sign the informed consent document, can communicate with the Investigator, and can understand and comply with the requirements of the protocol.
10. Women of childbearing potential must have a negative serum or urine beta-human chorionic gonadotropin test within 72 hours prior to first dose of study drug to rule out pregnancy.
11. All men and women must agree to practice effective contraception during the entire study period and after discontinuing study drug, unless documentation of infertility exists.

    1. Sexually active, fertile women must use 2 effective forms of contraception (abstinence, intrauterine device, oral contraceptive, or double barrier device) from the time of informed consent until at least 6 months after discontinuing study drug.
    2. Sexually active men and their sexual partners must use effective contraceptive methods from the time of subject informed consent until at least 3 months after discontinuing study drug.

Exclusion Criteria:

1. The subject was diagnosed with acute promyelocytic leukemia.
2. The subject is receiving concomitant therapy that includes other chemotherapy that is or may be active against AML except for agents such as hydroxyurea, just to control the WBC count until chemotherapy or prophylaxis and/or treatment of opportunistic or other infection with antibiotics, antifungals, and/or antiviral agents, including therapy for meningeal disease (i.e., intrathecal chemotherapy), supportive measures, and medications as per standard of care up to Day 1 of L-Annamycin administration.
3. The subject received prior mediastinal radiotherapy.
4. The subject has central nervous system involvement.
5. The subject has any condition that, in the opinion of the Investigator, places the subject at unacceptable risk if he/she were to participate in the study.
6. The subject has an LVEF <50%, valvular heart disease, or severe hypertension. Cardiac subjects with a New York Heart Association classification of 3 or 4 will be excluded. (Cardiology consultation should be requested if any question arises about cardiac function). This also includes subjects with baseline QT/QTc interval >480 msec, a history of additional risk factors for torsade des pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome), and use of concomitant medications that significantly prolong the QT/QTc interval.
7. The subject has clinically relevant serious comorbid medical conditions including, but not limited to, active infection, recent (less than or equal to 6 months) myocardial infarction, unstable angina, symptomatic congestive heart failure, uncontrolled hypertension, uncontrolled cardiac arrhythmias, chronic obstructive or chronic restrictive pulmonary disease, known positive status for human immunodeficiency virus and/or active hepatitis B or C, cirrhosis, or psychiatric illness/social situations that would limit compliance with study requirements.

   a. Subjects with a documented COVID diagnosis within 14 days of screening must have a documented negative PCR test and remain asymptomatic for 14 days from that test result before starting study medication.
8. The subject is pregnant, lactating, or not using adequate contraception.
9. The subject has a known allergy to anthracyclines and/or hypersensitivity to cytarabine, its excipients, or to any contrast media needed for imaging required per protocol.
10. The subject has any evidence of mucositis/stomatitis at the time of study entry or previous history of severe (≥Grade 3) mucositis from prior therapy.
11. The subject is required to use moderate or strong inhibitors and inducers of Cytochrome P450 family of enzymes (CYP) and transporters that cannot be held for 3 days prior to Day 1 and during treatment days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and identify the MTD/RP2D of L-Annamycin in combination with a standard regimen of cytarabine (Ara-C, cytosine arabinoside) | Day 1 through Day 28
  The number of patients who experience dose-limiting toxicities (DLT) will be captured at each dose level of LAnnamycin in order to determine the MTD/RP2D

SECONDARY OUTCOMES:
Pharmacokinetics - Area under the plasma concentration | Pre-dose and at 0.25, 0.5, 1, 2, 4, 8,12 and 24 hours after the start of liposomal annamycin infusion on Day 1 and Day 3
  Area under the plasma concentration - time curve (AUC) of annamycin and its metabolite, annamycinol, and of cytarabine, when administered.
Anti-leukemic activity | 15-35 Days after the start of therapy
  Determined by acute myeloid leukemia (AML) response rate based on the International Working Group (IWG) Response Criteria in AML (Cheson, 2003). Leukemia response rate will be evaluated by the investigator at the end of each L-Annamycin cycle based on bone marrow aspirate and peripheral blood evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram Dempke, MD, PhD, Study Director — Moleculin Biotech, Inc.
Locations (9):
- Italy (3):
  - Istituto Scientifico Romagolo per lo studio dei umori "Dino Amadori" (IRST) - IRCCS, Meldola, FC
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
- Poland (6):
  - Uniwersytecki Szpital Kliniczny Klinika Hematologii Nowotworow, Wroclaw, Dolnośląskie Województwo
  - SP ZOZ MsWiA z Warminsko-Mazurksim Centrum Onkologii w Olsztynie Oddzial Kliniczny Hematologii, Olsztyn, Warmian-Masurian Voivodeship
  - Apteka Szpitalna, Gdansk
  - Szpital Kliniczny Przemienienia Pańskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego, Poznan
  - Samodzielny Publiczny Szpital Kliniczny nr 1 im. Prof. Tadeusza Sokołowskiego w Szczecinie, Klinika Hematologii z Oddziałem Transplantacji Szpiku, Szczecin, Szczecin
  - Instytut Hematologii i Transfuzjologii, Klinika Hematologii, Warsaw, Warsaw